CLINICAL TRIAL: NCT01441973
Title: A Phase 2 Biomarker Study of Elotuzumab (Humanized Anti-CS1 Monoclonal IgG1 Antibody) Monotherapy to Assess the Association Between NK Cell Status and Efficacy in High Risk Smoldering Myeloma
Brief Title: Biomarker Study of Elotuzumab in High Risk Smoldering Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA204-011
Record Dates: First submitted 2011-09-27; First posted 2011-09-28 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elotuzumab, 20 mg/kg (Experimental): Intravenous solution administered in 28-day cycles. Cycle 1: Days 1 and 8. Cycle 2 and beyond: Day 1 only.
  Interventions: Biological: Elotuzumab (BMS-901608; HuLuc63)
- Elotuzumab, 10 mg/kg (Experimental): Intravenous solution administered in 28-day cycles. Cycle 1 and 2: Days 1, 8, 15, and 22. Cycle 3 and beyond: Days 1 and 15.
  Interventions: Biological: Elotuzumab (BMS-901608; HuLuc63)

INTERVENTIONS:
Biological: Elotuzumab (BMS-901608; HuLuc63)

SUMMARY:
The purpose of this study is to determine whether elotuzumab will improve response in patients with high risk smoldering myeloma who have more CD56^dim cells (a marker for the health of the body's immune system)

DETAILED DESCRIPTION:
Intervention model: Dosing is sequential

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Key Inclusion Criteria:

Participants with a confirmed diagnosis, according to criteria of the International Myeloma Working Group, of smoldering multiple myeloma, considered high risk according to the following:

* Serum monoclonal (M) protein ≥3 gm/dL and bone marrow plasma cells (BMPC) ≥10% or
* Serum M protein 1-3 g/dL and BMPC ≥10% and abnormal free light chain ratio of <0.125 or >8.0
* Urine M protein >200 mg/24 hours, ≥10% BMPC, and serum free light chain ratio ≤0.125 or ≥8.0

Key Exclusion Criteria:

* Active multiple myeloma
* Monoclonal gammopathy of undetermined significance
* Active plasma cell leukemia
* Positive for hepatitis B or C virus or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-12-28 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2017-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (12):
  - Sharp Clinical Oncology Research, San Diego, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Va Connecticut Healthcare System, West Haven, Connecticut
  - Winship Cancer Institute., Atlanta, Georgia
  - University Of Chicago Medical Center, Chicago, Illinois
  - Investigative Clinical Research Of Indiana, Llc, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School Of Medicine, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Mid Dakota Clinic, Pc, Bismarck, North Dakota

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled a total of 41 participants, and 31 received treatment. The 10 participants enrolled who did not receive treatment failed to meet the inclusion criteria.
Groups:
- Elotuzumab, 20 mg/kg: Participants in 2 arms were enrolled sequentially. The first group of participants received elotuzumab intravenously at a dose of 20 mg/kg on Days 1 and 8 per 28-day cycle for Cycle 1 and then on Day 1 only in subsequent cycles.
- Elotuzumab, 10 mg/kg: Participants in the second group received elotuzumab intravenously at a dose of 10 mg/kg weekly per 28-day cycle in Cycles 1 and 2, then on Days 1 and 15 in subsequent cycles.
Period: Overall Study
Arm/Group | Elotuzumab, 20 mg/kg | Elotuzumab, 10 mg/kg
Started | 15 | 16
Completed | 0 (Still receiving treatment) | 0 (Still receiving treatment)
Not Completed | 15 | 16
Not completed — Disease progression | 8 | 6
Not completed — Adverse event unrelated to study drug | 3 | 2
Not completed — Participant request to discontinue | 1 | 1
Not completed — Poor compliance/noncompliance | 0 | 1
Not completed — Administrative reason by sponsor | 3 | 5
Not completed — Participant withdrew consent | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Elotuzumab, 20 mg/kg | Elotuzumab, 10 mg/kg | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.0 (9.75) | 59.3 (9.37) | 59.2 (9.40)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 10 | 13 | 23
  65 years and older to younger than 75 years | 5 | 2 | 7
  75 years and older | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 14 | 15 | 29
  Black or African American | 1 | 1 | 2
Serum monoclonal (M) protein [Mean (Standard Deviation); unit: g/L] | 29.5 (15.19) | 21.9 (11.46) | 25.6 (13.72)
Urine M protein [Mean (Standard Deviation); unit: g/day] | 0.208 (0.6199) | 0.094 (0.2131) | 0.149 (0.4532)
Time from diagnosis to enrollment [Mean (Standard Deviation); unit: Months] | 31.75 (37.572) | 36.81 (35.103) | 34.37 (35.798)

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Who Died and With Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, and Infusion Reactions
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: From day of last patient, first dose to 6 months
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Groups:
- Elotuzumab, All Dosages: All participants on Elotuzumab therapy. Comprised of both the 20mg/kg and 10mg/kg arms
Arm/Group | Elotuzumab, 20 mg/kg | Elotuzumab, 10 mg/kg | Elotuzumab, All Dosages
Number analyzed (Participants) | 15 | 16 | 31
Participants
  Deaths | 0 | 0 | 0
  SAEs | 8 | 7 | 15
  AEs leading to discontinuation | 4 | 2 | 6
  Infusion reactions | 4 | 1 | 5

2. Primary Outcome: Linear Regression of Maximal Percent Reduction in Serum Monoclonal (M) Protein on Baseline Percent CD56^Dim Cells in Bone Marrow
Description: Estimated using linear regression model, with baseline CD56^dim cells as the independent covariate, and maximal percent reduction in serum M protein as the dependent variable. For 1 patient who had nonmeasurable disease at baseline, the percent change in serum kappa-lambda difference was used instead of the percent change in serum M protein. Unit of measure=percent change from baseline in M protein cells/ percent change in CD56^dim cells (% chg from BL in M pro/% chg CD56^dim cs)
Time Frame: From day of last patient, first dose to 6 months
Population: All participants who received at least 1 dose of study drug and had the required data (4 participants did not have baseline data available).
Measure: Number (95% Confidence Interval); unit: % chg from BL in M pro/% chg CD56^dim cs
Arm/Group | Elotuzumab, 20 mg/kg | Elotuzumab, 10 mg/kg | Elotuzumab, All Dosages
Number analyzed (Participants) | 13 | 12 | 31
% chg from BL in M pro/% chg CD56^dim cs | -2.562 [-5.439 to 0.316] | 2.464 [0.086 to 4.842] | 0.274 [-1.722 to 2.270]

3. Secondary Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Grade 3-4 Abnormality
Description: Clinical laboratory evaluations included hematology, chemistry, and liver and renal functioning.
Time Frame: From date of first dose to date of last dose plus 60 days (assessed up to August 2017, approximately 59 months
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Elotuzumab, 20 mg/kg | Elotuzumab, 10 mg/kg | Elotuzumab, All Dosages
Number analyzed (Participants) | 15 | 16 | 22
Participants
  Lymphocytes | 2 | 1 | 3
  Hyponatremia | 1 | 1 | 2
  Hyperkalemia | 0 | 1 | 1
  Hyperglycemia | 1 | 2 | 3

4. Secondary Outcome: Number of Participants With a Dose- or Concentration-related Effect on QTcF Interval, PR Interval, QRS Interval, and Heart Rate
Description: All on-treatment electrocardiograms (ECGs) were performed in triplicates ( 1 ECG test equaled 3 consecutive individual 12-lead ECGs performed within a 4-minute period). The timing of the ECG was critical to the endpoint of the study. The investigative site documented any deviations from the protocol or procedures related to ECG collection or serum sampling. No ECGs were excluded due to timing deviations; no deviations were considered clinically relevant and all ECG data were included.
Time Frame: cycle 1 to first day of cycle 3 assessed up to 08/17, approximately 59 months
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Elotuzumab, 20 mg/kg | Elotuzumab, 10 mg/kg | Elotuzumab, All Dosages
Number analyzed (Participants) | 15 | 16 | 31
Participants | 0 | 0 | 0

5. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: The probability was estimated from the K-M curve of subjects being alive and without disease progression (modified IMWG criteria) at 2 years from the initiation of study therapy by dose cohort
Time Frame: Up to 2 years from the initiation of study therapy by dose cohort (approximately 24 months)
Population: All treated participants
Measure: Number (90% Confidence Interval); unit: Probability of Progression Free Survival
Arm/Group | Elotuzumab, 20 mg/kg | Elotuzumab, 10 mg/kg | Elotuzumab, All Dosages
Number analyzed (Participants) | 15 | 16 | 31
Probability of Progression Free Survival | 0.71 [0.45 to 0.86] | 0.54 [0.31 to 0.72] | 0.62 [0.45 to 0.75]

6. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the number of participants with stringent compete response [SCR], complete response [CR], very good partial response [VGPR], and partial response [PR])/number of participants in arm, expressed as a percentage. Confidence intervals computed using the Clopper and Pearson method. SCR=CR plus normal free light chain ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence. CR=Negative immunofixation on serum and urine and 5% or fewer plasma cells in bone marrow. VGPR=Serum and urine monoclonal (M) protein detectable by immunofixation but not on electrophoresis or 90% reduction in serum M protein level plus urine M protein level <100 mg/24 hour. PR=50% reduction of serum M protein and reduction in 24-hour urinary M protein by 90% or to <200 mg/24 hour
Time Frame: From first dose to date of progression or objective response (assessed up to August 2017, approximately 59 months)
Population: All treated participants
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Elotuzumab, 20 mg/kg | Elotuzumab, 10 mg/kg | Elotuzumab, All Dosages
Number analyzed (Participants) | 15 | 16 | 31
Percentage of participants | 13.3 [2.4 to 36.3] | 6.3 [0.3 to 26.4] | 9.7 [2.7 to 23.2]

ADVERSE EVENTS:
Arm/Group | Elotuzumab(E) : 10 mg/kg/Dose | Elotuzumab(E) : 20 mg/kg/Dose
Serious Adverse Events (participants affected / at risk) | 7/16 | 8/15
Other Adverse Events (participants affected / at risk) | 16/16 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elotuzumab(E) : 10 mg/kg/Dose (N=16) | Elotuzumab(E) : 20 mg/kg/Dose (N=15)
Vertigo (Ear and labyrinth disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elotuzumab(E) : 10 mg/kg/Dose (N=16) | Elotuzumab(E) : 20 mg/kg/Dose (N=15)
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 1
Blepharitis (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 0
Eye discharge (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 2 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Photopsia (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 1 | 0
Retinal disorder (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 4
Dental discomfort (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Gingival pain (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 3
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Oral disorder (Gastrointestinal disorders) | 1 | 0
Palatal disorder (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1
Tongue blistering (Gastrointestinal disorders) | 1 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Catheter site pain (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 2 | 4
Chronic fatigue syndrome (General disorders) | 0 | 1
Cyst (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1
Fatigue (General disorders) | 10 | 8
Feeling cold (General disorders) | 2 | 0
Feeling jittery (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 3
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 4 | 2
Pain (General disorders) | 2 | 1
Peripheral swelling (General disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Ocular icterus (Hepatobiliary disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 2
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Ear infection viral (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 2 | 1
Herpes zoster (Infections and infestations) | 0 | 3
Hordeolum (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Lyme disease (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 3
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Purulence (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 5 | 2
Sinusitis (Infections and infestations) | 3 | 1
Sinusitis bacterial (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 12 | 9
Urinary tract infection (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood calcium increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 1
Eosinophil count increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Heart rate decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 1 | 0
Protein total increased (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 4
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 1 | 1
Muscle tone disorder (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 3
Paraesthesia (Nervous system disorders) | 4 | 1
Sciatica (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 7 | 3
Restlessness (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Testicular disorder (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Flushing (Vascular disorders) | 1 | 2
Haematoma (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.